CLINICAL TRIAL: NCT00517374
Title: A Multi-Centre Clinical Study in Spinal Cord Injury Patients in Mainland China and Hong Kong
Status: Completed | Type: Observational
Sponsor: China Spinal Cord Injury Network (Network)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Director, Clinical Trial Centre, The University of Hong Kong
Other Study IDs: CN100
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To establish a solid foundation, e.g. a network and a coordinating centre for testing new SCI therapies in forthcoming randomised controlled multi-centre clinical trials following international standards and guidelines.

DETAILED DESCRIPTION:
This is a multicentre, observational, registry study of outcome data on SCI patients in Mainland China and Hong Kong. The target population consists of patients who have a SCI, where acute SCI is defined as <7 days post-injury and chronic SCI is defined as >12 months post-initial SCI surgery.

A total of 600 patients (300 acute and 300 chronic) will be enrolled from 6 cities in Mainland China (namely: Beijing, Shanghai, Guangzhou, NingBo, Xi'an and Kunming) and Hong Kong. The duration of the study will be one year, with a total of 4 visits.

ELIGIBILITY:
Inclusion Criteria:

General

1. Male or female adult subjects, 18 to 65 years of age
2. Have a clinical diagnosis of SCI, defined by MRI
3. Voluntarily signs and dates an Informed Consent Form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to any study-specific procedures

   Acute SCI Study Group:
4. Has an acute SCI (defined as < 7 days post-injury)

Chronic SCI Study Group:

4. Has a chronic SCI (defined as > 12 months post-initial SCI surgery)

Exclusion Criteria:

General

1. Severe head injury
2. Is medically or mentally unstable according to the judgement of the Investigator
3. History of Multiple Sclerosis or peripheral demyelinating disease
4. Likely to have experimental therapy
5. Any criteria, which, in the opinion of the investigator, suggests that the subject would not be compliant with the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each study enrolled Hospital in China and Hong Kong is expected to recruit 20 chronic spinal cord injury patients, who have never had any cell therapy treatment for spinal cord injur before.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2005-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wise Young, MD, PhD, Study Director — Unaffilated
Locations (17):
- China (17):
  - First Affiliated Hospital of Medical College, Shantou University, Shantou, Guangdong
  - Ningbo Second People Hospital, Ningbo, Zhejiang
  - Beijing Army General Hospital, Beijing
  - Beijing University People's Hospital, Beijing
  - Beijing Xishan Hospital, Beijing
  - China Rehabilitation Research Center, Beijing
  - Nanfang Hospital, Guangzhou
  - Second Affliliated Hospital of Sun Yat-sen University, Guangzhou
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Chengdu Army Kuming General Hospital, Kunming
  - Changhai Hospital, Shanghai
  - Shanghai East Hospital, Shanghai
  - Zhongshan Hospital, Shanghai
  - Tianjin Medical University Hospital, Tianjin
  - Xian Jiaotong University Second Hospital, Xi'an
  - Xijing Hospital, Xi'an